CLINICAL TRIAL: NCT04382508
Title: Coronavirus Infection in Primary or Secondary Immunosuppressed Children and Adults.
Acronym: ImmunoCOVID
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Alder Hey Children's NHS Foundation Trust (Other); Birmingham Children's Hospital (Other); Bradford Royal Infirmary (Other); Bristol Royal Hospital for Children (Other); Cardiff and Vale University Health Board (Other Government); Great North Children's Hospital (Unknown); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Leeds Teaching Hospitals NHS Trust (Unknown); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Nottingham Children's Hospital (Unknown); Royal Alexandra Children's Hospital (Other); Royal Hospital for Sick Children, Glasgow (Unknown); Royal Manchester Children's Hospital (Unknown); Royal Marsden NHS Foundation Trust (Other); Northern Care Alliance NHS Group (Other); Royal Sussex County Hospital (Other); Sheffield Children's NHS Foundation Trust (Other); St George's University Hospital National Health Service Foundation Trust (Unknown); Swansea Bay University Health Board (Other); University College London Hospitals (Other); University Hospitals Coventry and Warwickshire National Health Service Trust (Unknown); East Lancashire Hospitals National Health Service Trust (Unknown); Imperial College Healthcare National Health Service Trust (Unknown); National Heatlh Service Ayrshire and Arran (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHM CHI1061
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-03

CONDITIONS: Immune Suppression; Immune Deficiency; Infection; COVID; Children, Adult
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — A weekly questionnaire will be filled in

SUMMARY:
A weekly questionnaire is sent to patients and parents of patients who are vulnerable for infections. Possible symptoms of COVID19 are asked for and use of healthcare services and testing for COVID19. Weekly reports are being send to the national institutions to update advice given to this group.

DETAILED DESCRIPTION:
This study is designed to allow immunosuppressed children, their parents or adult patients to self-record their experiences of COVID-19 and other viral respiratory illnesses. Patients, parents and of immunosuppressed patients and patients aged 16-17 yrs will be provided with online information and asked to fill in online questionnaires at baseline and weekly thereafter. Information collected includes medication, symptoms, contact with health care providers, test results and impact on daily activities. Data will be collected and analysed weekly to be able to monitor any potential risk factors for severe disease. This study is complementary to, and not overlapping with, the global ISARIC World Health Organisation protocol that will be studying COVID-19 cases admitted to all National Health Service (NHS) Trusts, including all children.

ELIGIBILITY:
Inclusion Criteria:

* Children part: Parent of immunosuppressed patient aged <16 years or immunosuppressed patient aged 16-17 years
* Adult part: Immunosuppressed patient aged >17 years
* Family or themselves able to complete the questionnaire which will be in English (due to current resources available translation will not be possible)
* Reliable access to the internet

Exclusion Criteria:

* Unable to understand English

Age Groups: Child, Adult, Older Adult
Study Population: Children and adults vulnerable for infection due to a condition or to medication they are using.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-03-22 (Actual); Primary Completion 2021-03-21 (Estimated); Study Completion 2021-03-21 (Estimated)

PRIMARY OUTCOMES:
To describe COVID19 infection in children/adults who are vulnerable for infection in an outpatients setting | 1 year
  To describe frequency of cough, fever, diarrhoea, shortness of breath, sore throat, blocked nose, red eyes, headache, joint pain, muscle pain, fatigue, chills, nausea, vomiting, diarrhoea over a year

SECONDARY OUTCOMES:
Number of children/adults tested positive for COVID19 | 1 year
  Patient/parent reported positive tests for COVID19
Number of children/adults admitted in hospital because of COVID19 | 1 year
  Patient/parent reported admissions in hospital because of COVID19
To assess the impact of COVID19 infection on the daily activities of immunosuppressed adults and children | 1 year
  Patient/parent reported effect of COVID19 on daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Hans de Graaf, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS FT, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaunak M, Patel R, Driessens C, Mills L, Leahy A, Gbesemete D, Owens DR, Lucas JS, Faust SN, de Graaf H; ImmunoCOVID19 study group. COVID-19 symptom surveillance in immunocompromised children and young people in the UK: a prospective observational cohort study. BMJ Open. 2021 Mar 17;11(3):e044899. doi: 10.1136/bmjopen-2020-044899. PMID 33737439
- See also: Study website — https://www.uhs.nhs.uk/ClinicalResearchinSouthampton/Public-and-patients/Featured-research-studies/Featured-research-ImmunoCOVID19-study.aspx